CLINICAL TRIAL: NCT00920998
Title: A Pharmacokinetics Study to Evaluate the Effect of Food Intake on PK Profile of Z-338 in Healthy Volunteers
Brief Title: Effect of Food Intake on Pharmacokinetic Profiles of Z-338
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 443-CL-503
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Z-338; YM443; healthy volunteers
MeSH Terms: interventions — Z 338

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. Z-338 (Experimental): 3-way cross-over study (drug administration 3-times in fasted and 2 fed conditions)
  Interventions: Drug: Z-338

INTERVENTIONS:
Drug: Z-338 — oral
  Other Names: YM443

SUMMARY:
To evaluate the effects of food intake on plasma concentration of Z-338 in healthy volunteers.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the influence of food intake on the pharmacokinetic profiles of Z-338 in healthy volunteers by a 3-way cross-over method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Body weight: 50.0 - 80.0 kg
* BMI: 17.6 - 26.4

Exclusion Criteria:

* Receiving an investigational new drug within 120 days of the study
* Receiving medical treatment drugs within 7 days of the study
* Blood donation before the study

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Z-338 | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan